CLINICAL TRIAL: NCT07008157
Title: Efficacy of a Multimodal Conservative Rehabilitation Program for Bladder Control in Individuals With Incomplete Spinal Cord Injury: A Randomized Controlled Trial
Brief Title: Rehabilitation Program for Bladder Control in Individuals With Incomplete Spinal Cord Injury
Acronym: BCSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT.BU.EC.18
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
Keywords: Rehabilitation Program; Bladder Control; Incomplete Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: both participants and outcome assessors blinded to group assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): received IFC, PFMT, motor MIT, and timed voiding (TV)1. IFC interferential current, pelvic floor muscles training, timed voiding, and motor imagery training
  Interventions: Other: 1. IFC; Other: 2. Timed voiding.; Other: motor imagery training; Other: pelvic floor muscles training
- control group (Active Comparator): participants received interferential current therapy, timed voiding, and pelvic floor muscles training
  Interventions: Other: 1. IFC; Other: 2. Timed voiding.; Other: pelvic floor muscles training

INTERVENTIONS:
Other: 1. IFC — IFC therapy was applied while the patient lay in a supine position with the knees slightly apart. Each treatment session involved four electrodes enclosed in lint cloth covers. Two electrodes were positioned bilaterally on the lower abdomen, just below the anterior superior iliac spines (ASIS), while the remaining two were placed on the inner surfaces of both thighs. To maintain hygienic standards, the cloth covers were replaced for each participant at every session. The intervention was administered three times weekly over an eight-week period. A frequency range of 0-10 Hz was used, and the current intensity was carefully adjusted based on each patient's comfort and tolerance. Each IFC session lasted 15 minutes, with the aim of modulating pelvic region activity to support improved bladder function. This protocol was implemented three times per week over an eight-week period
Other: 2. Timed voiding. — The approach involved instructing participants to follow a fixed, scheduled voiding routine, typically every 3 hours, irrespective of the sensation to urinate. Additionally, patients were advised to adjust their toileting posture by sitting and leaning forward at an angle of approximately 45 degrees, allowing adequate time for complete bladder emptying. The technique also included practicing double voiding, where the individual would stand up and sit down again after the initial void to help ensure maximum bladder evacuation
Other: motor imagery training — Prior to initiating MIT, participants watched a 10-minute instructional video in a quiet treatment space, illustrating proper PFM contractions through both visual and auditory cues. The therapist provided a detailed explanation, using a simple analogy of the bladder as a balloon filled with urine, connected by a tube (the urethra) to the outside, and controlled by the PFM. It was explained that contracting these muscles tightens the balloon, holding back urine, whereas weak or relaxed muscles may lead to leakage. Patients were then guided to mentally visualize contracting and holding these muscles until they reached a suitable time and place (the toilet), without physically performing the action. Following this explanation, patients were asked to sit comfortably with their eyes closed and spend 10 minutes visualizing the movement and control of their PFM while remaining physically relaxed. Throughout the session, the therapist used open-ended prompts to help maintain the patient's focu
  Arms: experimental group
Other: pelvic floor muscles training — Before beginning each treatment session, participants were instructed to empty their bladders to promote comfort and relaxation during the exercises. All patients were taught a structured PFMT routine, to be performed daily in multiple positions such as lying, sitting, and standing. The program consisted of contracting the PFM for 10 seconds, followed by a 10-second relaxation period, with this sequence repeated 15 times in each session. To gradually enhance the endurance of the slow-twitch muscle fibers, both contraction and relaxation times were increased by one second each week. In addition, to activate and strengthen the fast-twitch muscle fibers, patients were directed to perform 20 quick, repetitive contractions and relaxations of the levator ani muscles - simulating the act of stopping urine flow, followed by a 10-second rest. This rapid contraction sequence was repeated for 2 to 4 sets in each session. This protocol was implemented three times per week over an eight-week period

SUMMARY:
This prospective, randomized, double-blind clinical trial (with both participants and outcome assessors blinded to group assignments) was carried out at the outpatient clinic of the Faculty of Physical Therapy, Cairo University, following patient referrals. Participants were recruited between October 2024 and April 2025 from the National Institute of Urology and Nephrology in Mataria, as well as the Department of Urology and Nephrology at Kasr Alaini Hospital. All diagnoses were verified by a consultant urologist. The study received ethical approval from the Institutional Review Board of the Faculty of Physical Therapy, Benha University, Egypt, and written informed consent was obtained from each participant prior to enrollment.

Participants Individuals between 18 and 65 years of age presenting with OAB symptoms, confirmed through urodynamic testing, and diagnosed with ISCI classified as AIS C or D above the L1 spinal level, were considered eligible for inclusion in this study. Participants were required to be medically stable, able to follow study protocols, and willing to provide informed consent. Exclusion criteria included those with complete spinal cord injury (AIS A), current urinary tract infections, a history of pelvic malignancy, prior bladder or pelvic surgeries, or significant cognitive or psychiatric disorders.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind clinical trial (with both participants and outcome assessors blinded to group assignments) was carried out at the outpatient clinic of the Faculty of Physical Therapy, Cairo University, following patient referrals. Participants were recruited between October 2024 and April 2025 from the National Institute of Urology and Nephrology in Mataria, as well as the Department of Urology and Nephrology at Kasr Alaini Hospital. All diagnoses were verified by a consultant urologist. The study received ethical approval from the Institutional Review Board of the Faculty of Physical Therapy, Benha University, Egypt, and written informed consent was obtained from each participant prior to enrollment.

Participants Individuals between 18 and 65 years of age presenting with OAB symptoms, confirmed through urodynamic testing, and diagnosed with ISCI classified as AIS C or D above the L1 spinal level, were considered eligible for inclusion in this study. Participants were required to be medically stable, able to follow study protocols, and willing to provide informed consent. Exclusion criteria included those with complete spinal cord injury (AIS A), current urinary tract infections, a history of pelvic malignancy, prior bladder or pelvic surgeries, or significant cognitive or psychiatric disorders. Simple randomization was applied to allocate participants into one of two groups: the EG, which received IFC, PFMT, motor MIT, and timed voiding (TV); and the CG, which received IFC, PFMT, and TV. The randomization process involved a computer-generated sequence created using dedicated software to ensure an equal number of participants in each group. Allocation concealment was maintained by placing group assignments in sealed, opaque envelopes, which were opened sequentially as participants were enrolled in the study.

Outcome Measures

1. Urodynamic assessments
2. The International Consultation on Incontinence Questionnaire - Short Form (ICIQ-UI SF)
3. PFM strength Treatment procedures

1. IFC therapy 2. Timed voiding. 3. Motor imagery Training 4. PFMT

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 65 years of age

  * presenting with OAB symptoms
  * diagnosed with ISCI classified as AIS C or D above the L1 spinal level

Exclusion Criteria:

* complete spinal cord injury
* current urinary tract infections
* a history of pelvic malignancy
* prior bladder or pelvic surgeries
* significant cognitive or psychiatric disorders

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
1. Urodynamic assessments | at three time points: baseline, after 8 weeks of treatment, and at an 8-week follow-up
  These evaluations were carried out by experienced clinicians to maintain consistency and accuracy, providing real-time measurements of bladder function in a controlled environment. The procedure involved positioning the patient either supine or seated, followed by the insertion of a sterile catheter through the urethra into the bladder for fluid instillation and pressure monitoring. During cystometric testing, the bladder was gradually filled with sterile saline at a steady rate, while intravesical and abdominal pressures were continuously recorded. Key parameters measured included MCC, LPP, and the bladder volume at the first sensation of the urge to void
Body Mass Index | baseline, after 8 weeks of treatment, and at an 8-week follow-up.
  In this study, Body Mass Index (BMI) was used as an anthropometric measure to assess the weight status of patients with incomplete spinal cord injuries. BMI was calculated using the formula: BMI = weight (kg) / height² (m²). The classification of BMI values followed the guidelines established by the World Health Organization, where individuals with a BMI less than 18.5 kg/m² were considered underweight, those between 18.5-24.9 kg/m² were classified as having a normal weight, values from 25.0-29.9 kg/m² indicated overweight, and a BMI of 30.0 kg/m² or higher was categorized as obesity (World Health Organization, 2000).

SECONDARY OUTCOMES:
2. The International Consultation on Incontinence Questionnaire - Short Form (ICIQ-UI SF) | at three time points: baseline, after 8 weeks of intervention, and at an 8-week follow-up
  ICIQ-UI SF is a widely recognized, validated, and reliable tool designed to assess the severity of urinary incontinence and its effect on QOL. It has demonstrated strong validity and reliability, producing consistent, reproducible results across diverse clinical and research populations (Avery et al., 2004). In the present study, the ICIQ-UI SF was administered at three time points: baseline, after 8 weeks of intervention, and at an 8-week follow-up, in accordance with the study's schedule for evaluating changes in urinary symptoms and related QOL

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available when required

REFERENCES:
- [Background] Elfahl AM, Abd El Baky AM, Yousef MT, Elgohary HM. High Versus Low Frequency Transcutaneous Electric Nerve Stimulation On Chronic Venous Lower Limb Ulceration Randomized Controlled Trial. Int J Low Extrem Wounds. 2025 Jun;24(2):376-382. doi: 10.1177/15347346221093860. Epub 2022 Apr 14. PMID 35422171
- See also: Related Info — https://orcid.org/0000-0001-5531-1875